CLINICAL TRIAL: NCT04794582
Title: Prevention of Incisional Hernia After Renal Transplantation Using ProGrip Mesh
Brief Title: Prevention of Incisional Hernia After Renal Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Victoria Gómez Dos Santos, Head of Renal Surgery and Transplantation Section, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 445/20
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Incisional Hernia; Kidney Transplantation; Postoperative Complications
Keywords: Incisional Hernia; Kidney Transplantation
MeSH Terms: conditions — Incisional Hernia; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Blinded parallel randomized clinical trial. A stratified allocation by the variable obesity will be performed using permuted blocks of variable size in each stratum. To guarantee the concealment of the randomization sequence, the randomization codes will be kept in opaque envelopes with correlative numerical identification that will be opened once it has been verified that the patient meets the inclusion criteria and has signed the informed consent form.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For observer masking, the observer (outcomes assessor) will belong to the General Surgery team that is not directly involved with the transplantation procedure and agrees not to verify the assignment in the transplantation surgical protocol.
  Finally, the masking of the analyst (investigator) is achieved through collaboration with the Clinical Biostatistics Unit in the data analysis of the study (independent analyst) using a pseudo-anonymized database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ProGrip® Mesh reinforcement (Active Comparator): Once the closure has been completed in 2 muscle-aponeurotic planes with continuous synthetic suture (Monomax® USP 0), the closure will be completed by placing the ProGrip® macroporous polypropylene monofilament mesh in supra-aponeurotic position using the surface with the polylactic acid microgrips, which act as Velcro, in direct contact with the superficial aponeurotic plane constituted by the aponeuroses of the greater oblique muscle and the crescentic line of the anterior rectus abdominis muscle. The polylactic acid microgrips provide immediate fixation, making additional fixation with stitches unnecessary, which makes the technique very easy to use and systematize among the different surgeons of the transplant team. The procedure is completed with the placement of a low caliber round Jackson-Pratt subcutaneous drain (10F) connected to a vacuum system that will be removed on post-transplant day 2 or 3
  Interventions: Device: ProGrip™ Self-Gripping Polyester Mesh
- Monomax® USP 0 2 planes closure (No Intervention): The control group will proceed according to standard clinical practice with closure using the technique in 2 muscle-aponeurotic planes with very long-term (3 months) absorbable synthetic continuous suture of poly(4-hydroxybutyrate), monofilament, elastic (Monomax® USP 0) according to the small-bites technique. In order to achieve masking of the participating subject, a small-bore (10F) Jackson-Pratt drain connected to a vacuum system will be placed in the subcutaneous space at the end of the procedure in a manner similar to the intervention group. In both treatment groups, the subcutaneous drain will be removed on post-transplant day 2 or 3.

INTERVENTIONS:
Device: ProGrip™ Self-Gripping Polyester Mesh — Supra-aponeurotic placement of ProGrip® macroporous polyester mesh in the supra-aponeurotic position
  Arms: ProGrip® Mesh reinforcement

SUMMARY:
Randomized clinical trial to determine the efficacy of mesh reinforcement in laparotomy closure in renal transplantation as measured by reduction in the incidence of incisional hernia at 2 years post-transplantation.

DETAILED DESCRIPTION:
As defined by the European Hernia Society, eventration or incisional hernia is any defect in the abdominal wall with or without an associated bulge in the area of a surgical scar that is noticeable or palpable by physical examination or imaging tests. Incisional hernias after abdominal organ transplantation are of special interest since transplant recipients undergo immunosuppressive treatment that may increase the risk of developing incisional hernias due to their impact on the healing process. It is estimated that the incidence of incisional hernia after renal transplantation ranges from 1.6 to 18% and increases to 1.7-32.4% and 13.0-34.8% after liver and pancreatic transplantation respectively. Incisional hernias are a major source of morbidity and most require surgical repair at some point in time. Regarding patient-related factors, female sex and obesity have been identified as potential risk factors. In the case of immunosuppressive medication, nucleotide synthesis inhibitors such as mycophenolate and m-TOR inhibitors such as sirolimus have been associated with a higher incidence of incisional hernia. With regard to factors specifically related to the surgical wound, surgical wound infection and type of incision have been identified as risk factors. In 2018 Simson et al published a systematic review of the existing literature that highlights the limited scientific evidence that is primarily made up of case series review. We conducted a retrospective observational study that identified an incidence of 12.5% of incisional hernia on physical examination, which increase to 29.8% on radiological examination (CT) with a median time to diagnosis of 17.1 months (2.5 - 23.9). An additional 17.5% of muscle atrophy was observed.

To determine the efficacy of mesh reinforcement in laparotomy closure in renal transplantation as measured by reduction in the incidence of incisional hernia at 2 years post-transplantation a randomized clinical trial is proposed.

In accordance with the extensive experience and recommendations of the Abdominal Wall Section of the General and Digestive Surgery Department of our hospital, we intend to carry out a randomized clinical trial for the prophylactic use of Medtronic ProGrip™ Self-Gripping Polyester Mesh mesh reinforcement in supra-aponeurotic position. This mesh features polylactic acid (PLA) microgrips that act as Velcro, providing immediate, strong and uniform fixation, weighing 82 g/m2 before PLA resorption and 41 g/m2 after resorption (low density). The use of this mesh combines the effectiveness demonstrated by the macropore meshes in the treatment of incisional hernias, a high simplicity of use provided by its capacity for self-fixation for which it is equipped with the so-called absorbable microgrips of polylactic acid that adhere quickly and easily to the underlying tissue and safety. This mesh has proven its usefulness and safety for the prophylaxis of eventration in patients with other types of lateral incisions.

Patients in ProGrip group will be treated with self-gripping polyester and Polylactic acid meshes providing a sutureless fixation.

In the control group, closure will be performed according to standard clinical practice using the technique in 2 muscle-aponeurotic planes with very long-term (3 months) absorbable synthetic continuous suture of poly(4-hydroxybutyrate), monofilament, elastic (Monomax® USP 0) according to the small-bites technique.

Study participation will start at signature of informed consent and each patient will be assessed before surgery. A close follow-up will be performed at 3, 6, 12 months (clinical visit, physical examination, laboratory tests, adverse effects), and final evaluation at 24 months (clinical visit, physical examination, laboratory tests, adverse effects and radiological examination -CT-) after surgery, which will end the participation to the study.

160 adult (>18 years) recipients of a first kidney transplantation divided in 2 groups will be included in the study. Allocation by the obesity variable, which is a determinant risk factor in the response to the intervention, will be carried out using permuted blocks of variable size in each stratum.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for first kidney transplant

Exclusion Criteria:

* Patient receiving a second or successive renal transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of mesh reinforcement in laparotomy closure in renal transplantation measured by radiological diagnosis (CT) | 24 months
  To determine the efficacy of mesh reinforcement in laparotomy closure in renal transplantation measured by radiological diagnosis (CT) of incisional hernia at 2 years post-transplantation.

SECONDARY OUTCOMES:
To determine the safety of mesh reinforcement in laparotomy closure in renal transplantation | 3, 6, 12 and 24 months
  To determine the safety of mesh reinforcement in laparotomy closure in renal transplantation measured by determining the incidence of surgical wound complications: number of seromas, number of surgical wound infections, incidence and severity of acute and chronic pain, and need for mesh removal.

OTHER OUTCOMES:
To determine the efficacy of mesh reinforcement in laparotomy closure in renal transplantation as measured by the reduction in the incidence of incisional hernia at 2 years post-transplantation measured by radiological diagnosis (CT) | 24 months
  Reduction in the incidence of incisional hernia at 2 years post-transplantation.
To determine the incidence of incisional hernia surgery in post-renal transplantation measured by physical examination at 3, 6 and 12 months and by radiological diagnosis (CT) at 24 months | 3, 6, 12 and 24 months
  To determine the incidence of incisional hernia surgery in post-renal transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: VICTORIA GOMEZ, Principal Investigator — Fundación para la Investigación Biomédica del Hospital Unive
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data collected in the project will be recorded and stored in an electronic data capture tool developed for this project under REDCap (Research Electronic Data Capture, Vanderbilt University, TN, USA) that complies with national and international regulatory and legal requirements, including GDPR Regulation (EU) 2016/679. Data generated will be uploaded to provide access to the PI. Data will be shared by the PI only with the research team members. Access data security would be granted and supervised by the Data Protection Officer (DPO). All patient level data will be accessed only in coded and anonymized form.
  Once the objectives of the project have been achieved, the data used will be deposited in the internal REDCap repository of IRYCIS, which is the Institutional Repository of the Ramón y Cajal Health Research Institute. Access to the internal repository data for other researchers who may be legitimately interested in them will be subject to the approval of an ethics commission.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the end of the study for 6 months
Access Criteria: After approval of an specific ethics commission

REFERENCES:
- [Derived] Gomez-Dos-Santos V, Lopez-Plaza JA, Molina-Villar JM, Blazquez-Hernando L, Diez-Nicolas V, Jimenez-Cidre M, Porrero-Guerrero B, Rodriguez-Patron R, Arias-Funez F, Muriel-Garcia A, Fernandez-Cebrian JM, Burgos-Revilla FJ. Prevention of incisional hernia after kidney transplantation: study protocol for a randomized controlled trial. Trials. 2023 Aug 14;24(1):528. doi: 10.1186/s13063-023-07545-0. PMID 37580782